CLINICAL TRIAL: NCT00963495
Title: Phase 1 Study Evaluating the Tolerance and Biological Activity of Oral Clioquinol in Patients With Relapsed or Refractory Hematological Malignancy
Brief Title: Study Evaluating the Tolerance and Biological Activity of Oral Clioquinol in Patients With Relapsed or Refractory Hematological Malignancy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADS1.0
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Myelodysplasia; Lymphoma, Non-Hodgkin; Hodgkin's Lymphoma; Multiple Myeloma
Keywords: clioquinol; relapsed and refractory hematologic malignancy; ALL; HD; CLL; High risk myelodysplasia (MDS) with an IPSS score >2.5; CML blast crisis; Relapsed or refractory acute myeloid leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Recurrence; Hematologic Neoplasms | interventions — Clioquinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clioquinol (Experimental): Patients will take Clioquniol at various doses depending on which dose level they come into the study at. Once a MTD has been determined, the new patients that enter into the trial will then take it at that level.
  Interventions: Drug: Clioquinol

INTERVENTIONS:
Drug: Clioquinol — Patients will take Clioquniol at escalating doses depending on when they enter into the trial.

SUMMARY:
This is an open-label, single arm phase 1 study to evaluate the dose-limiting toxicity, maximum tolerated dose, and recommended phase II dose of Clioquinol in patients with relapsed or refractory hematologic malignancies. The study will also characterize Cliquinol's safety, tolerability and pharmacodynamic effect.

DETAILED DESCRIPTION:
This is an open-label, single arm study. Approximately 4-48 patients will be enrolled. Patients will receive 800mg/day of Clioquinol at the start of the trial and the dose will be increased by 800mg with each subsequent level until the MTD is determined. Patients will then increase their frequency of the drug. Response to Clioquinol will be determined on day 21 for the 8 and 15 day dosing schedule and on day 28 for the 22 day dosing schedule ( 1 cycle). Patients who have demonstrated a response to the drug will be eligible to receive up to 5 additional cycles at the same dose and frequency every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), high risk myelodysplasia (MDS) with an IPSS score > 2.5, Non-Hodgkin's lymphoma (NHL), Hodgkin's lymphoma (HD) or multiple myeloma, for which all potentially curative or standard salvage therapy options have been exhausted.
2. ECOG performance status < 2.
3. Biochemical values within the following range:

   * Serum creatinine < 2x upper limit of normal.
   * Total bilirubin < 2x upper limit of normal, AST and ALT < 5x upper limit of normal.
   * Normal serum B12 level.
4. Ability to maintain adequate oral intake of medication.
5. Ability to understand and sign informed consent.
6. Toxicity from prior chemotherapy has resolved.

Exclusion Criteria:

1. Uncontrolled systemic infection.
2. Uncontrolled intracurrent illness.
3. Pregnant or breast feeding.
4. CNS disease.
5. Neurologic symptoms related to intracurrent illnesses or unexplained causes.
6. Psychiatric illness that would limit compliance with study.
7. Receiving other systemic chemotherapy, other than hydroxyurea to control circulating blast counts, within 10 days of study entry. Hydroxyurea is permitted, however the dose must be stable and unchanged in the 7 days prior to initiation with Clioquinol.
8. Prior therapy with Clioquinol.
9. Use of other investigational antileukemic therapy within two weeks of study entry.
10. Given the neurological side of Clioquinol in the Japanese population, this population, this trial will exclude patients who have a parent of Oriental or Japanese origin or who self-identify as Oriental or Japanese (Appendix 9.2).
11. Active ocular problems including visual migraines and glaucoma.
12. Use of oral or intravenous heavy metal supplements including copper, zinc, and nickel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the dose-limiting toxicity (DLT), maximum tolerated dose, and recommended phase II dose. To partially characterize the pharmacokinetics of Clioquinol in plasma following single and multiple oral dosing. | Varies

SECONDARY OUTCOMES:
To determine the pharmacodynamic effects of Clioquinol on activity of the proteasome and relationship to the steady-state plasma concentrations of Cliquinol following multiple dosing, and to determine the response rate of Cliquinol. | Varies

CONTACTS AND LOCATIONS:
Overall Officials: Mark Minden, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada